CLINICAL TRIAL: NCT03916471
Title: Comparison of Efficacy and Side Effects Between the Obtryx and Solyx Band With 5-year Follow-up. Prospective, Randomized and Non-inferiority Study
Brief Title: Comparison of Efficacy and Side Effects Between the Obtryx and Solyx Band With 5-year Follow-up.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOSTON2018
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S (SOLYX) (Experimental): The Solyx™SIS System is an innovative mid-urethral sling single incision system consisting of a 9 cm long polypropylene mesh, whose mid-urethral portion (4 cm) is detanged to potentially resist deformation and to reduce irritation to the urethral wall. Snap-fit to delivery device tip allows for advanced placement control and, therefore, the tensioning through the forward and reverse functions performed with this delivery device.
  Interventions: Device: Solyx™ SIS System
- O (OBTRYX II) (Experimental): The Obtryx II System (Halo) is a transobturator sling designed to allow inter-operative adjustability with minimal tissue disruption. It consists of two delivery devices (one patient right and one patient left) and one mesh assembly. The mesh assembly is comprised of a polypropylene knitted mesh with dilator legs and a center tab. At the distal ends of the dilator legs there are association loops designed to be placed in the needle slot of the distal end of the delivery device. The disposable delivery device consists of a handle with a stainless steel needle. The needle is designed to facilitate the passage of the mesh assembly through bodily tissues for placement through the obturator foramen.
  Interventions: Device: Obtryx™ II System (Halo)

INTERVENTIONS:
Device: Solyx™ SIS System — Single-incision sling system
  Arms: S (SOLYX)
Device: Obtryx™ II System (Halo) — Transobturator Mid-urethral Sling System
  Arms: O (OBTRYX II)

SUMMARY:
Boston2018 post-market clinical study is a prospective, randomized, non-inferiority study to assess the efficacy and adverse events of the Solyx™ Single Incision Sling (SIS) System compared to the gold-standard Obtryx™ II Sling System, in patients with stress urinary incontinence (SUI) and long-term follow-up (5 years).

DETAILED DESCRIPTION:
Randomized prospective non-inferiority study, in which we evaluate patients with stress urinary incontinence (SUI) who undergo surgical treatment consisting of a minimal incision in the suburethral area of the vaginal mucosa for a mesh insertion in order to:

Main Objective:

To compare the continence rate (objective) between Solyx and Obtryx II meshes in patients with SUI. This rate will be determined by an effort test.

Secondary Objectives:

* To compare the continence rate (subjective) between both meshes.
* To compare variations in Pad-Test.
* To asses patient satisfaction.
* To evaluate both techniques regarding quality and sexual life modifications.
* To compare both techniques regarding early complications (up to 30 days post implantation).
* To compare the appearance and persistence of late complications (from 30 days onwards).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with symptomatic stress urinary incontinence candidates for stress-free bands
* Age > or = 40 years
* informed consent signed by the patient

Exclusion Criteria:

* patients who are pregnant or wish to become
* patients who need anticoagulant
* active vaginal or urinary infection
* previous surgical interventions for the treatment of incontinence
* body mass index > 35

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female diagnosed with symtomatic stress urinary incontinence
Enrollment: 166 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Continence rate (Objective) assessed by an effort test | Month 1
  For the analysis of the objective cure of incontinence, an effort test will be carried out through three strokes of cough, with bladder volume between 200-300 ml in a lithotomy position.
Continence rate (Objective) assessed by an effort test | Month 6
  For the analysis of the objective cure of incontinence, an effort test will be carried out through three strokes of cough, with bladder volume between 200-300 ml in a lithotomy position.
Continence rate (Objective) assessed by an effort test | Year 1
  For the analysis of the objective cure of incontinence, an effort test will be carried out through three strokes of cough, with bladder volume between 200-300 ml in a lithotomy position.
Continence rate (Objective) assessed by an effort test | Year 2
  For the analysis of the objective cure of incontinence, an effort test will be carried out through three strokes of cough, with bladder volume between 200-300 ml in a lithotomy position.
Continence rate (Objective) assessed by an effort test | Year 3
  For the analysis of the objective cure of incontinence, an effort test will be carried out through three strokes of cough, with bladder volume between 200-300 ml in a lithotomy position.
Continence rate (Objective) assessed by an effort test | Year 4
  For the analysis of the objective cure of incontinence, an effort test will be carried out through three strokes of cough, with bladder volume between 200-300 ml in a lithotomy position.
Continence rate (Objective) assessed by an effort test | Year 5
  For the analysis of the objective cure of incontinence, an effort test will be carried out through three strokes of cough, with bladder volume between 200-300 ml in a lithotomy position.

SECONDARY OUTCOMES:
Continence rate (Subjective) assessed by Incontinence Questionnaire-Urinary Short Form (ICQ-SF) | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  Incontinence Questionnaire-Urinary Short Form (ICQ-SF): continent patient when the reduction is equal to or greater than 50% of the value prior to the intervention.
Pad test | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  1 hour pad test: After a spontaneous urination the patient will place a compress that will be weighed previously.
  After, the patient has to drink a half liter of water in 15 minutes sitting. Between the minute 15 to 45 has to walk and / or go up / down stairs. From minute 45-60 the patient has to get up and sit 10 times, cough 10 times, run 1 minute, lift an object from the ground 10 times and washes his/her hands 1 minute.
  According to the difference in weight of the compress, it will be cataloged as follows:
  ≤ 1 gram -> continent. 1.1-9.9 grams -> mild incontinence. 10-49.9 grams -> moderate incontinence. > 50 grams -> severe incontinence
Patient satisfaction assessed by PGI-I (Patient Global Impression of Improvement) | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  PGI-I consider a patient satisfied when the patient answer " better or much better".
Patient satisfaction assessed by the "Global Satisfaction Test" | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  Global satisfaction assessment will be required, with a rank 1-5, being 1 very satisfied and 5 very dissatisfied.
Patient satisfaction assessed by the "Recommendations questionnarie" | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  The recommendation grade will be assessed through the question "will you recommend this surgical treatment for other patients?", the possible answer are Yes or No.
Evaluation of life quality improvement assessed by I-QoL questionnaire (Urinary Incontinence-Specific Quality of Life Instrument) | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  To assess the life quality impact, I-QoL questionnaire (Urinary Incontinence-Specific Quality of Life Instrument) will be used , this questionnaire, is composed by 22 items. The highest punctuation mean better life quality. The modification of 2.5 points, which has been considered in this questionnaire, is the minimum clinically significant modification in patients presenting SUI. This questionnaire is validated in Spanish.
Evaluation of sexual life, assessed by PSIQ 12 questionnaire (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire ) | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  To assess the impact on sexual life, the PSIQ 12 questionnaire (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire ) will be used. It is composed of 12 items graded from "never" to "always". This questionnaire is validated in heterosexual women who have urinary incontinence and / or pelvic organ prolapse. Scores are calculated for each item with a value of "always = 0" and for "never = 4". It is used inversely in items 1-4.
Early complications assessed by Post-Mictional Residue | Day 0, 7-10 days after the intervention, Month 1
  Are considered by the urgency of urination, the inability to void, the presence of PMR greater than 50% of the total volume after spontaneous voiding or the presence of pain that prevents ambulation, in the first 30 days after the intervention.
  For the elevated PMR assessment, perineal ultrasound measurement will be carried out after spontaneous micturition. If the PMR measurement will be higher or equal, probing would be performed to obtain the exact residue. If it is pathological, proceed according to the usual practice.
Early complications assessed by OAB-q questionnaire (Overactive Bladder symptom and health-related quality of life questionnaire) | Day 0, 7-10 days after the intervention, Month 1
  OAB-q questionnaire (Overactive Bladder symptom and health-related quality of life questionnaire). Individual answer punctuation: lowest 0, highest 5 .If the score ≥8 will proceed according to the usual practice.
Long term complications assessed by OAB-q questionnaire (Overactive Bladder symptom and health-related quality of life questionnaire) | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  OAB-q questionnaire (Overactive Bladder symptom and health-related quality of life questionnaire). Individual answer punctuation: lowest 0, highest 5 .If the score ≥8 will proceed according to the usual practice.
Early complications assessed by VAS (Visual Analogue Scale) | Day 0, 7-10 days after the intervention, Month 1
  Only when the patient has a pain that prevents ambulation. VAS: Pain scale for quantification of pain. Range 0 to 10. 0: No pain 5: Distressing pain 10: Unbearable pain
Long term complications assessed by "Extrusion" (integrity of the vaginal mucus) | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  Extrusion: The integrity of the vaginal mucus will be checked in all the visits that are made. If there is evidence of mesh extrusion, it is classified as asymptomatic / symptomatic and according to its size (greater or less than 1 cm).
Long term complications assessed by emergence of recurrent urinary tract infections (UTIs) | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  Urinary tract infection: in the presence of at least 1 monthly urinary tract infections (UTI), the patient will be considered to have developed repeat UTIs.
Long term complications assessed by "Emptying dysfunction" | Month 1, month 6, year 1, year 2, year 3, year 4 and year 5.
  Persistent urinary retention at 30 days will be considered as a long term complication.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Garcia, Principal Investigator — Instituto de Investigación y Politécnico La Fe
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thom DH, Nygaard IE, Calhoun EA. Urologic diseases in America project: urinary incontinence in women-national trends in hospitalizations, office visits, treatment and economic impact. J Urol. 2005 Apr;173(4):1295-301. doi: 10.1097/01.ju.0000155679.77895.cb. PMID 15758785
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Ulmsten U, Henriksson L, Johnson P, Varhos G. An ambulatory surgical procedure under local anesthesia for treatment of female urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):81-5; discussion 85-6. doi: 10.1007/BF01902378. PMID 8798092
- [Background] Ward KL, Hilton P; UK and Ireland TVT Trial Group. Tension-free vaginal tape versus colposuspension for primary urodynamic stress incontinence: 5-year follow up. BJOG. 2008 Jan;115(2):226-33. doi: 10.1111/j.1471-0528.2007.01548.x. Epub 2007 Oct 25. PMID 17970791
- [Background] Nilsson CG, Palva K, Rezapour M, Falconer C. Eleven years prospective follow-up of the tension-free vaginal tape procedure for treatment of stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Aug;19(8):1043-7. doi: 10.1007/s00192-008-0666-z. Epub 2008 Jun 6. PMID 18535753
- [Background] Nambiar A, Cody JD, Jeffery ST, Aluko P. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2017 Jul 26;7(7):CD008709. doi: 10.1002/14651858.CD008709.pub3. PMID 28746980
- [Background] Ford AA, Rogerson L, Cody JD, Ogah J. Mid-urethral sling operations for stress urinary incontinence in women. Cochrane Database Syst Rev. 2015 Jul 1;(7):CD006375. doi: 10.1002/14651858.CD006375.pub3. PMID 26130017
- [Background] Ford AA, Rogerson L, Cody JD, Aluko P, Ogah JA. Mid-urethral sling operations for stress urinary incontinence in women. Cochrane Database Syst Rev. 2017 Jul 31;7(7):CD006375. doi: 10.1002/14651858.CD006375.pub4. PMID 28756647
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839